CLINICAL TRIAL: NCT06033989
Title: Clinical and Radiographic Evaluation of the Effect of Hyaluronic Acid Surface Treatment Versus Sandblasted Acid Etched Surface Treatment on Stability of Delayed Dental Implant in Posterior Maxilla. Comparative Randomized Clinical Trial (RCT).
Brief Title: Clinical and Radiographic Evaluation of the Effect of Hyaluronic Acid Surface Treatment Versus Sandblasted Acid Etched on Stability of Delayed Dental Implant in Posterior Maxilla.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shihanah Yousef Ahmed Alkashi, Master's degree candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Shihanah1993
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Missing Teeth; Bone Loss
Keywords: Dental implant; Stability; Osseointegration; Hyaluronic acid; Sandblasted acid etched
MeSH Terms: conditions — Anodontia; Bone Diseases, Metabolic | interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyaluronic acids (Experimental): Hyaluronic acid has a huge potential to speed up the healing process and increase implant stability by enhancing bone/implant interaction and new bone formation.
  Interventions: Drug: Hyaluronic acid; Procedure: Delayed dental implant
- Sandblasting acid etched (Active Comparator): Sandblasting and acid etching is the most commonly used basic method for modifying the surface of dental implants . the sandblasting procedure "roughs up" the outer layer of the implant , creating a surface that is easier for the bone to grip as the implant heals.
  Interventions: Drug: sandblasted, and acid-etched; Procedure: Delayed dental implant

INTERVENTIONS:
Drug: Hyaluronic acid — Delayed dental implant placement after application of surface treatment to enhance Osseointegration and healing .
  Arms: Hyaluronic acids
Drug: sandblasted, and acid-etched — Delayed dental implant placement after application of surface treatment to enhance Osseointegration and healing .
  Arms: Sandblasting acid etched
Procedure: Delayed dental implant — Surgical procedure of delayed dental implant in posterior maxilla after application of surface treatment to enhance Osseointegration and healing .

SUMMARY:
Clinical and Radiographic Evaluation of the Effect of Hyaluronic Acid Surface Treatment Versus Sandblasted Acid Etched on Stability of Delayed Dental Implant in Posterior Maxilla.

DETAILED DESCRIPTION:
A dental implant is one of the procedures to restore missing teeth , to achieved the stability for implant success is the direct growth of bone to the implant surface, known as Osseointegration.As a result, bone stability around dental implants is determined by factors that the implantologist may or may not directly influence, such as local bone quality and bone metabolism, as well as systemic factors such as age, systematic chronic diseases and lifestyle (e.g., smoking habits).Treatment-related factors include augmentation material, implant design (macro and micro), surgical procedures, and loading protocols. Therefore , it may be needed for a surface treatment could alter the topography, chemical content, and roughness of the surface and result in various biological reactions. The surface treatment can also increase the area of contact between the implant and the supporting bone . The rationale is evaluate Increasing the implant stability around implants placed by using hyaluronic acid that act to improving the connection between implant and bone .Sandblasting and acid etching is the most commonly used basic method for modifying the surface of dental implants . the sandblasting procedure "roughs up" the outer layer of the implant,creating a surface that is easier for the bone to grip as the implant heals.While hyaluronic acid and its derivatives have a strong chance of osseointegration and mineralization and have been utilized extensively for bone repair.

ELIGIBILITY:
Inclusion Criteria:

* Patients with missing teeth in posterior maxilla.
* Both genders males and females will be included.
* Age from 18-60 years.

Exclusion Criteria:

* General contraindications to implant surgery.
* Subjected to irradiation in the head and neck area less than 1 year before implantation.
* Untreated periodontitis.
* Poor oral hygiene and motivation.
* Uncontrolled diabetes.
* Pregnant or nursing.
* Substance abuse.
* Psychiatric problems or unrealistic expectations.
* Severe bruxism or clenching.
* Immunosuppressed or immunocompromised.
* Treated or under treatment with intravenous amino-bisphosphonates.
* Active infection or severe inflammation in the area intended for implant placement.
* Unable to open mouth sufficiently to accommodate the surgical tooling.
* Patients participating in other studies, if the present protocol could not be properly followed.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Implant stability | 0-3 months
  It is assessed by using Osstell To determine the stability after intervention scale from 60 to 70 ISQ 60 low stability 70 high stability .

SECONDARY OUTCOMES:
soft tissue healing | 10 days
  It is assessed by using gingival index in Clinical examination scale from 0 Normal 1 Mild inflammation 2 Moderate inflammation 3 Severe inflammation .
bone density | 3 months
  It is assessed by using CBCT To determine the density of bone after intervention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peck MT, Marnewick J, Stephen L. Alveolar ridge preservation using leukocyte and platelet-rich fibrin: a report of a case. Case Rep Dent. 2011;2011:345048. doi: 10.1155/2011/345048. Epub 2011 Jul 3. PMID 22567435
- [Background] Meredith N. Assessment of implant stability as a prognostic determinant. Int J Prosthodont. 1998 Sep-Oct;11(5):491-501. PMID 9922740
- [Background] Velasco-Ortega E, Jimenez-Guerra A, Monsalve-Guil L, Ortiz-Garcia I, Nicolas-Silvente AI, Segura-Egea JJ, Lopez-Lopez J. Long-Term Clinical Outcomes of Treatment with Dental Implants with Acid Etched Surface. Materials (Basel). 2020 Mar 27;13(7):1553. doi: 10.3390/ma13071553. PMID 32230917
- [Background] Massaro C, Rotolo P, De Riccardis F, Milella E, Napoli A, Wieland M, Textor M, Spencer ND, Brunette DM. Comparative investigation of the surface properties of commercial titanium dental implants. Part I: chemical composition. J Mater Sci Mater Med. 2002 Jun;13(6):535-48. doi: 10.1023/a:1015170625506. PMID 15348583
- [Background] Cervino G, Meto A, Fiorillo L, Odorici A, Meto A, D'Amico C, Oteri G, Cicciu M. Surface Treatment of the Dental Implant with Hyaluronic Acid: An Overview of Recent Data. Int J Environ Res Public Health. 2021 Apr 27;18(9):4670. doi: 10.3390/ijerph18094670. PMID 33925742
- [Result] Gupta R, Gupta N, Weber, DDS KK. Dental Implants. 2023 Aug 8. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470448/ PMID 29262027